CLINICAL TRIAL: NCT06251778
Title: NatiOnal Referral cenTEr Study of Transthyretin Amyloid Cardiomyopathy(ATTR) Patients on Tafamidis: Real World Prospective Study
Brief Title: NatiOnal Referral cenTEr Study of Transthyretin Amyloid Cardiomyopathy(ATTR) Patients on Tafamidis
Acronym: NOTE-ATTR
Status: Recruiting | Type: Observational
Sponsor: Paolo Milani (Other)
Responsible Party: Sponsor-Investigator, Paolo Milani, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Organization: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Other Study IDs: AC-022-IT
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Amyloidosis; Amyloidosis Cardiac; ATTR Amyloidosis Wild Type
MeSH Terms: conditions — Amyloidosis; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All ATTRwt patients on tafamidis 61 mg treatment will be clinically evaluated before treatment initiation and subsequently every six months for the eligibility to continue tafamidis treatment, according to Italian Medicines Agency regulations. C onsidering the significant risk of developing heart rhythm disturbances due to cardiac amyloidosis, especially in transthyretin form (ATTRwt), in routine clinical practice a stricter heart rhythm monitoring is recommended in ATTRwt patients. Moreover, particular attention is usually paid for those who present atrio-ventricular and/or intraventricular block at the baseline electrocardiogram. Data about rhythm disturbances and diuretic dose need will be collected during the planned physical examination every six months and the Holter ECG monitoring requested by the physician at the end of every planned clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ATTRwt amyloidosis.
* 18 years or older;
* evidence of cardiac involvement at echocardiography or cardiac MRI.
* No known prior history of atrial fibrillation or major bradyarrhythmia (second degree atrioventricular block, third-degree atrioventricular block, high-grade atrioventricular block or alternating right and left branch block)
* female patients who are postmenopausal for at least 1 year before the screening visit
* patients on therapy or candidates for therapy with tafamidis 61 mg
* voluntary written consent must be given before performance of any study-related procedure not part of standard medical care with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

* Non-ATTR amyloidosis;
* NYHA class III and IV;
* Pregnant or nursing women;
* Previous pacemaker implantation;
* any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with a fully comprehension of the written consent form

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of ATTRwt disease and eligible for tafamidis treatment according to the national drug regulatory agency criteria and no prior history of atrial trachy-arrhythmia and/or bradyarrhythmias in their past medical history will undergo screening procedure to be enrolled in the present study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-01-26 (Estimated); Study Completion 2026-01-26 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of atrial tachy-arrhythmia and brady-arrhythmias requiring pacemaker and/or defibrillator | 18 months
  All ATTRwt patients eligible for tafamidis with no prior history of atrial tachy-arrhythmia or brady-arrhythmias will be prospectively enrolled. The events (arrythmias incidence) will be collected by the usually rhythm monitoring that physician will recommend at the end of clinical evaluation according to clinical practice

SECONDARY OUTCOMES:
patient diuretic dose need (i.e. Furosemide), reported as mg/Kg/die | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No